CLINICAL TRIAL: NCT01741207
Title: Evaluation of N-acetylcystein on Biomarkers of Platelet Activation , Cardiac Necrosis and Coronary Reperfusion in Patients Undergoing Percutaneous Coronary Intervention
Brief Title: Effect of N-acetylcystein in Myocardial Infarction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 524; IRCT201210118698N2 (Registry Identifier: IRCT)
Record Dates: First submitted 2012-11-30; First posted 2012-12-04 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-11

CONDITIONS: Acute Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): control This group is without N-acetylcystein : just receives standard treatment
- N-acetylcystein (Active Comparator): receive N-acetylcystein in addition to standard treatment Ampoule 200 mg/ml
  Interventions: Drug: N-acetylcystein

INTERVENTIONS:
Drug: N-acetylcystein — Active Comparator: N-acetylcystein receive N-acetylcystein in addition to standard treatment
  Other Names: EXI-NACE,NAC
  Arms: N-acetylcystein

SUMMARY:
We designed this study to evaluate the effect of N-acetylcystein on biomarkers of platelet activation , cardiac necrosis and coronary reperfusion in patients undergoing percutaneous coronary intervention.

DETAILED DESCRIPTION:
Percutaneous coronary intervention(PCI) is one of the standard therapies for acute coronary syndrome. Despite major advances in PCI procedure, impaired myocardial perfusion frequently occurred after primary PCI and resulted in a larger infarct size and increased morbidity and mortality.Reperfusion injury process can be resulted in additional death of cardiomyocytes and it is suggested that oxidative stress is a contributing factor to induce reperfusion injury.During PCI,trauma occurs to the arterial endothelium, causes the activation and aggregation of platelets.

It is estimated that approximately 25% of patients undergoing PCI have significant postprocedural creatinine kinase (CK)/creatinine kinase myocardial band (CK-MB) elevations and approximately 50% of patients have significant post-procedural troponin elevations. The most common complication of PCI is a cell damage to cardiomyocyte that can be diagnosed by postprocedure elevation of cardiac markers. N-acetylcystein have several positive effect on platelet and vascular function and infarct size.

This study is a randomized clinical trial (RCT) evaluating the effect of N-acetylcystein on biomarkers of platelet activation and coronary reperfusion in patients undergoing percutaneous coronary intervention. Double blind randomized clinical trial on 100 patients in 2 groups (intervention & control) is conducted. Patients with confirmed ST-elevation myocardial infarction included in this study. Patients were excluded if they had: emergency for cardiac bypass; cardiogenic shock and rescue percutaneous coronary intervention. Patients in Intervention group were administered 100 mg/kg Iv bolus N-acetylcystein and then 480mg intracoronary and 10mg/kg/h over 12 hours after percutaneous coronary intervention and patients in control group received standard regimens. Primary outcome was platelet activation biomarkers assessment before and 24 hours after percutaneous coronary intervention and secondary outcome was effect of N-acetylcystein on CK-MB and high sensitive Troponin T, 6 and 12 hours after percutaneous coronary intervention.Patients were assessed for coronary blood flow after percutaneous coronary intervention with the use of TIMI flow and myocardial blush grade.

Major adverse cardiac events (MACE) will be evaluated as a secondary endpoint after 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Myocardial infarction patients who were candidate of primary PCI

Exclusion Criteria:

* Rescue PCI
* Emergency for cardiac bypass
* Cardiogenic shock
* Life expectancy less than 6 months
* Age less than 18 years old
* Uncontrolled hypertension
* Thrombocytopenia
* Malformation or aneurysm
* Sever chronic kidney disease
* Sever liver failure
* Major surgery within 3 months
* Unsatisfactory to enter the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Biomarkers of platelet activation (P selectin- CD40L-IL[Interleukin] 10- TGF[Transforming Growth Factor]-beta) | Change from the baseline after 24 hours

SECONDARY OUTCOMES:
Cardiac Necrosis Biomarkers (CKMB, Troponin T) | Change from the baseline after 12 hours
  difference between study and control group in 6 and 12 hrs after percutaneous coronary intervention
score of coronary blood flow(TIMI flow and MBG) | Change from the baseline after percutaneous coronary intervention
MACE (Major Adverse Cardiac Effect) | 30 days
  Defined as Need for Target Revascularization, Myocardial Infarction and Death

CONTACTS AND LOCATIONS:
Overall Officials: Azita Hajhossein Talasaz, PharmD,BCPS, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- Teran Heart Center, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Nozari Y, Eshraghi A, Talasaz AH, Bahremand M, Salamzadeh J, Salarifar M, Pourhosseini H, Jalali A, Mortazavi SH. Protection from Reperfusion Injury with Intracoronary N-Acetylcysteine in Patients with STEMI Undergoing Primary Percutaneous Coronary Intervention in a Cardiac Tertiary Center. Am J Cardiovasc Drugs. 2018 Jun;18(3):213-221. doi: 10.1007/s40256-017-0258-8. PMID 29322434